CLINICAL TRIAL: NCT01463072
Title: Efficacy and Tolerability of Nanoparticle Albumin Bound Paclitaxel (Abraxane) in Patients 65 and Older With Locally Advanced or Metastatic Breast Cancer
Brief Title: Nab-Paclitaxel in Treating Older Patients With Locally Advanced or Metastatic Breast Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11139; NCI-2011-03295 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 118196; 124494; 11139 (Other: City of Hope Comprehensive Cancer Center); P30CA033572 (NIH)
Record Dates: First submitted 2011-10-25; First posted 2011-11-01 (Estimated); Results first posted 2022-07-26 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Locally Advanced Breast Carcinoma; Metastatic Breast Carcinoma; Recurrent Breast Carcinoma; Stage III Breast Cancer AJCC v7; Stage IIIA Breast Cancer AJCC v7; Stage IIIB Breast Cancer AJCC v7; Stage IIIC Breast Cancer AJCC v7; Stage IV Breast Cancer AJCC v6 and v7
MeSH Terms: conditions — Breast Neoplasms | interventions — 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (nab-paclitaxel) (Experimental): Patients receive nab-paclitaxel IV over 30 minutes on days 1, 8, and 15. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Nab-paclitaxel; Other: Questionnaire Administration

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Nab-paclitaxel — Given IV
  Other Names: ABI 007; ABI-007; Abraxane; Albumin-bound Paclitaxel; Albumin-Stabilized Nanoparticle Paclitaxel; Nanoparticle Albumin-bound Paclitaxel; Nanoparticle Paclitaxel; Paclitaxel Albumin; paclitaxel albumin-stabilized nanoparticle formulation; protein-bound paclitaxel
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial studies the side effects of nab-paclitaxel in treating older patients with breast cancer that has spread from where it started to nearby tissue or lymph nodes (locally advanced) or to other places in the body (metastatic). Drugs used in chemotherapy, such as nab-paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the tolerability (grade 2-5 toxicity, neuropathy grade 2 or higher, need for dose reductions, or delays) of weekly nab-paclitaxel in older adults with locally advanced or metastatic breast cancer.

SECONDARY OBJECTIVES:

I. To evaluate the efficacy (response and time to progression) of weekly nab-paclitaxel in older adults with locally advanced or metastatic breast cancer using a stratification factor based on patient age (at least 5 patients age 75 years or older and no more than 15 patients age 65-70 years).

II. To explore predictors of the need for dose reduction, dose delays, or grade 2-5 toxicity and neuropathy grade 2 or higher based on a cancer-specific geriatric assessment.

OUTLINE:

Patients receive nab-paclitaxel intravenously (IV) over 30 minutes on days 1, 8, and 15. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced or metastatic breast cancer
* Any estrogen receptor (ER), progesterone receptor (PR), or human epidermal growth factor receptor 2 (Her2neu) status as long as the patient will receive nab-paclitaxel alone
* First or second line chemotherapy treatment for metastatic disease
* Karnofsky performance status (KPS) >= 70%
* Resolution of grade >= 2 toxicity from prior therapy (other than alopecia)
* Peripheral neuropathy =< grade 1
* Absolute neutrophil count >= 1,500/mm^3
* Platelets >= 100,000 cells/mm^3
* Hemoglobin (Hb) >= 9.0 g/dl
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x institutional upper limit of normal
* Alkaline phosphatase =< 2.5 x upper limit of normal unless bone metastasis are present in the absence of liver metastases
* Bilirubin =< 1.5 mg/dl
* Creatinine clearance (calculated or 24 hour) >= 30 ml/min
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients may not be receiving any other investigational agents
* Untreated central nervous system (CNS) metastases or symptomatic CNS metastases requiring escalating doses of corticosteroids
* Known history of allergic reactions to paclitaxel
* Presence of any serious or uncontrolled infection
* Receipt of a taxane for adjuvant therapy or metastatic disease in the last 12 months

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-06-19 (Actual); Primary Completion 2017-05-17 (Actual); Study Completion 2026-05-18 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Mina Sedrak, Principal Investigator — City of Hope Medical Center
Locations (4):
- United States (4):
  - City of Hope medical, Duarte, California
  - City of Hope Antelope Valley, Lancaster, California
  - City of Hope South Pasadena, South Pasadena, California
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hurria A, Soto-Perez-de-Celis E, Blanchard S, Burhenn P, Yeon CH, Yuan Y, Li D, Katheria V, Waisman JR, Luu TH, Somlo G, Noonan AM, Lee T, Sudan N, Chung S, Rotter A, Arsenyan A, Levi A, Choi J, Rubalcava A, Morrison R, Mortimer JE. A Phase II Trial of Older Adults With Metastatic Breast Cancer Receiving nab-Paclitaxel: Melding the Fields of Geriatrics and Oncology. Clin Breast Cancer. 2019 Apr;19(2):89-96. doi: 10.1016/j.clbc.2018.10.002. Epub 2018 Oct 16. PMID 30503309

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Nab-paclitaxel)
Started | 40
Completed | 40
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Nab-paclitaxel)
Number analyzed (Participants) | 40
Age, Continuous [Mean (Full Range); unit: years] | 73 [65 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 33
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 29
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 40
Receptor status [Count of Participants; unit: Participants]
  HR-positive | 30
  Triple-negative | 10

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants With Grade 2-5 Toxicity Using National Cancer Institute Common Toxicity Criteria Version 4.0
Description: Will be graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. Rates and associated 95% exact Clopper and Pearson binomial confidence limits will be estimated for grade 2 or higher toxicities attributed to treatment.
Time Frame: During and after treatment, up to 2.5 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Nab-paclitaxel)
Number analyzed (Participants) | 40
percentage of participants | 90 [76 to 97]

2. Primary Outcome: Percent of Participants With Grade 3 or Higher Toxicities Attributable to Treatment
Description: Will be graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. Rates and associated 95% exact Clopper and Pearson binomial confidence limits will be estimated for grade 3 or higher toxicities attributed to treatment.
Time Frame: On treatment, 28 days per cycle up to 30 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Nab-paclitaxel)
Number analyzed (Participants) | 40
percentage of participants | 58 [41 to 73]

3. Primary Outcome: Rate of Participants With a Dose Reduction
Description: Rates and associated 95% exact Clopper and Pearson binomial confidence limits will be estimated for dose reduction.
Time Frame: On treatment, up to 30 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Nab-paclitaxel)
Number analyzed (Participants) | 40
percentage of participants | 50 [34 to 66]

4. Primary Outcome: Rate of Participants Requiring Dose Holds
Description: Rates and associated 95% exact Clopper and Pearson binomial confidence limits will be estimated for dose reduction.
Time Frame: While on treatment, up to 30 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Nab-paclitaxel)
Number analyzed (Participants) | 40
percentage of participants | 75 [59 to 87]

5. Secondary Outcome: Response Determined by Response Evaluation Criteria in Solid Tumors
Description: Rates and associated 95% exact Clopper and Pearson binomial confidence limits will be estimated for objective response rate (complete response [CR] + partial response [PR]).
  RECIST:
  Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes must have reduction in short axis to <10 mm
  Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters
  Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. Additionally, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered progression
  Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study
Time Frame: Up to 2.5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Nab-paclitaxel)
Number analyzed (Participants) | 40
Participants
  Complete remission | 1
  Partial remission | 13
  Stable disease | 16
  Progressive disease | 4
  Off treatment prior to disease assessment | 6
Statistical Analysis 1: Comparison: Treatment (Nab-paclitaxel); Test type: Other; Percent = 35, 95% CI 2-sided [21 to 52] — 35% of participants were responders (CR+PR)

6. Secondary Outcome: Median Progression Free Survival (PFS)
Description: PFS will be estimated using the product limit method of Kaplan and Meier.
Time Frame: From the date treatment begins until the first date on which recurrence, progression, or death due to any cause, assessed for about 1.5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Nab-paclitaxel)
Number analyzed (Participants) | 40
months | 6.5 [5.5 to NA] — Insufficient number of participants with events

7. Secondary Outcome: Cancer-specific Geriatric (CARG) Assessment
Description: General linear models and descriptive methods will be used to explore factors as identified by a CARG assessment that may be predictive of toxicity (grade 3 or higher adverse events) or dose reduction.
  The cancer specific geriatric assessment score includes an evaluation of functional status, co-morbidity, cognition, psychological stats, social functioning and support, and nutritional status. It assesses a patient's age, gender, height, weight, cancer type, dosage, number of chemotherapy agents, hemoglobin, hearing, number of falls in past 6 months, able to take own medicine, whether walking is limited, have physical or emotional problems interfered with social activities and serum creatinine.
  Scores can range from 0 to to 1, with a higher score indicating higher risk of chemotherapy toxicity. Scores from 0 to 5 are considered low risk, 6 to 9 are considered intermediate risk, and 10 to 19 are considered high risk.
Time Frame: CARG measured prior to treatment, toxicities and dose reduction measured up to 30 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Nab-paclitaxel)
Number analyzed (Participants) | 40
Participants
  Low CARG chemotherapy toxicity risk | 21
  Intermediate CARG chemotherapy toxicity risk | 15
  High CARG chemotherapy toxicity risk | 4
Statistical Analysis 1: Comparison: Treatment (Nab-paclitaxel); CARG chemotherapy toxicity risk predictive of chemotherapy toxicity (grade 3); Test type: Superiority; p = 0.01, Fisher Exact; Odds Ratio (OR) = 5.8, 95% CI 2-sided [1.3 to 33.1] — Ratio is intermediate/high toxicity risk over low toxicity risk
Statistical Analysis 2: Comparison: Treatment (Nab-paclitaxel); CARG chemotherapy toxicity risk predictive of dose reduction due to chemotherapy toxicity; Test type: Superiority; p = 0.02, t-test, 2 sided; Ratio of group means = 1.38, 95% CI 2-sided [1.04 to 1.80] — Ratio is dose reduction over no dose reduction

ADVERSE EVENTS:
Time Frame: On study, up to 2.5 years
Arm/Group | Treatment (Nab-paclitaxel)
All-Cause Mortality (participants affected / at risk) | 35/40
Serious Adverse Events (participants affected / at risk) | 14/40
Other Adverse Events (participants affected / at risk) | 40/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Nab-paclitaxel) (N=40)
Anemia (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Cardiac disorders - Other, specify (Cardiac disorders) | 1
Heart failure (Cardiac disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 2
Mucositis oral (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 4
Fatigue (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Allergic reaction (Immune system disorders) | 1
Urinary tract infection (Infections and infestations) | 1
Bronchial infection (Infections and infestations) | 1
Activated partial thromboplastin time prolonged (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Hyponatermia (Metabolism and nutrition disorders) | 1
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 1
Stroke (Nervous system disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Hematoma (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Nab-paclitaxel) (N=40)
Anemia (Blood and lymphatic system disorders) | 19
Conjunctivitis (Eye disorders) | 2
Diarrhea (Gastrointestinal disorders) | 4
Edema limbs (General disorders) | 2
Pain (General disorders) | 3
Fatigue (General disorders) | 23
Allergic reaction (Immune system disorders) | 2
Nail infection (Infections and infestations) | 2
Infections and infestations - Other, specify (Infections and infestations) | 3
Urinary tract infection (Infections and infestations) | 4
Skin infection (Infections and infestations) | 6
Upper respiratory infection (Infections and infestations) | 7
Aspartate aminotransferase increased (Investigations) | 2
Weight gain (Investigations) | 2
Lymphocyte count decreased (Investigations) | 8
Neutrophil count decreased (Investigations) | 17
White blood cell decreased (Investigations) | 25
Hyperglycemia (Metabolism and nutrition disorders) | 3
Hypokalemia (Metabolism and nutrition disorders) | 4
Dehydration (Metabolism and nutrition disorders) | 5
Hypocalcemia (Metabolism and nutrition disorders) | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Peripheral sensory neuropathy (Nervous system disorders) | 6
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Thromboembolic event (Vascular disorders) | 2
Hypotension (Vascular disorders) | 3
Hypertension (Vascular disorders) | 18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-23): https://cdn.clinicaltrials.gov/large-docs/72/NCT01463072/Prot_SAP_000.pdf